CLINICAL TRIAL: NCT05516641
Title: Do Prebiotics Change Intestinal Biome in Rectal Cancer Patients Undergoing Neoadjuvant Therapy
Brief Title: Prebiotics in Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2021.227
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer
Keywords: stage II; stage III; microbiome; prebiotic; racial disparities
MeSH Terms: conditions — Rectal Neoplasms | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prebiotic (Experimental): Soluble Corn Fiber
  Interventions: Dietary Supplement: Soluble Corn Fiber
- Control (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Soluble Corn Fiber — once daily additive to diet
  Arms: Prebiotic
Dietary Supplement: Maltodextrin — once daily additive to diet
  Arms: Control

SUMMARY:
A significant racial disparity in the incidence and mortality of CRC exists in the U.S. with African Americans having CRC incidence and mortality rates that are 20% and 40% higher than the general U.S. population. It has been demonstrated that the gut microbiome impacts tumor development and progression through multiple mechanisms, including impacting the tumoral immune response. However, it is unknown if microbiome modulating treatment can have an impact on CRC outcomes.

DETAILED DESCRIPTION:
A significant racial disparity in the incidence and mortality of CRC exists in the U.S. with African Americans having CRC incidence and mortality rates that are 20% and 40% higher than the general U.S. population. It has been demonstrated that the gut microbiome impacts tumor development and progression through multiple mechanisms, including impacting the tumoral immune response. However, it is unknown if microbiome modulating treatment can have an impact on CRC outcomes.

This is a pilot project to see if any changes are detected in stool and/or tissue samples in rectal cancer patients who receive a soluble corn fiber supplement during their neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Clinical diagnosis of stage 2 or stage 3 rectal cancer
3. Subjects who are women of child-bearing potential must not be pregnant or lactating
4. Have signed an approved informed consent form for the study
5. Be willing to comply with the protocol

Exclusion Criteria:

1. Patients with a cancer history (excluding the rectal cancer currently being addressed)
2. Allergic to corn or maltodextrin
3. Has, in the Investigator's opinion, any medical condition that makes the subject a poor candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Gut Flora modulation | 1 year
  fiber supplements with prebiotic effects modulate the gut and tumor associated microbiome leading to improved outcomes in stage II and III rectal cancer patients

SECONDARY OUTCOMES:
Microbiome changes | 6 months
  To characterize the changes in the gut and tumor associated microbiome
Immune Profile | 6 months
  To evaluate the impact of prebiotic fiber treatment and microbiome changes on the tumor immune profile known to be associated with favorable outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, PhD, Principal Investigator — Ochsner
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States